CLINICAL TRIAL: NCT05958979
Title: Effects of e-Cigarettes on Perceptions and Behavior - Remote Substudy # 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Adam Leventhal, Professor of Preventive Medicine, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Substudy #1: UP-20-00744
Record Dates: First submitted 2023-07-07; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Electronic Cigarette Use; Cigarette Smoking; Cigarette Use, Electronic; Vaping
Keywords: vaping; e-cigarette; vape; nicotine; tobacco
MeSH Terms: conditions — Vaping; Cigarette Smoking

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to use a varying number of e-liquids with differing marketing strategies.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (20):
- E-cigarette e-liquid 1 (Experimental)
  Interventions: Other: Control Marketing Strategies; Other: Experimental Marketing Strategies
- E-cigarette e-liquid 2 (Experimental)
  Interventions: Other: Control Marketing Strategies; Other: Experimental Marketing Strategies
- E-cigarette e-liquid 3 (Experimental)
  Interventions: Other: Control Marketing Strategies; Other: Experimental Marketing Strategies
- E-cigarette e-liquid 4 (Experimental)
  Interventions: Other: Control Marketing Strategies; Other: Experimental Marketing Strategies
- E-cigarette e-liquid 5 (Experimental)
  Interventions: Other: Control Marketing Strategies; Other: Experimental Marketing Strategies
- E-cigarette e-liquid 6 (Experimental)
  Interventions: Other: Control Marketing Strategies; Other: Experimental Marketing Strategies
- E-cigarette e-liquid 7 (Experimental)
  Interventions: Other: Control Marketing Strategies; Other: Experimental Marketing Strategies
- E-cigarette e-liquid 8 (Experimental)
  Interventions: Other: Control Marketing Strategies; Other: Experimental Marketing Strategies
- E-cigarette e-liquid 9 (Experimental)
  Interventions: Other: Control Marketing Strategies; Other: Experimental Marketing Strategies
- E-cigarette e-liquid 10 (Experimental)
  Interventions: Other: Control Marketing Strategies; Other: Experimental Marketing Strategies
- E-cigarette e-liquid 11 (Experimental)
  Interventions: Other: Control Marketing Strategies; Other: Experimental Marketing Strategies
- E-cigarette e-liquid 12 (Experimental)
  Interventions: Other: Control Marketing Strategies; Other: Experimental Marketing Strategies
- E-cigarette e-liquid 13 (Experimental)
  Interventions: Other: Control Marketing Strategies; Other: Experimental Marketing Strategies
- E-cigarette e-liquid 14 (Experimental)
  Interventions: Other: Control Marketing Strategies; Other: Experimental Marketing Strategies
- E-cigarette e-liquid 15 (Experimental)
  Interventions: Other: Control Marketing Strategies; Other: Experimental Marketing Strategies
- E-cigarette e-liquid 16 (Experimental)
  Interventions: Other: Control Marketing Strategies; Other: Experimental Marketing Strategies
- E-cigarette e-liquid 17 (Experimental)
  Interventions: Other: Control Marketing Strategies; Other: Experimental Marketing Strategies
- E-cigarette e-liquid 18 (Experimental)
  Interventions: Other: Control Marketing Strategies; Other: Experimental Marketing Strategies
- E-cigarette e-liquid 19 (Experimental)
  Interventions: Other: Control Marketing Strategies; Other: Experimental Marketing Strategies
- E-cigarette e-liquid 20 (Experimental)
  Interventions: Other: Control Marketing Strategies; Other: Experimental Marketing Strategies

INTERVENTIONS:
Other: Control Marketing Strategies — Participants will self-administer experimenter-provided e-cigarettes
Other: Experimental Marketing Strategies — Participants will self-administer experimenter-provided e-cigarettes

SUMMARY:
This study assess the ways in which e-cigarette product characteristics, such as marketing strategies, impact user experience to inform potential regulations.

DETAILED DESCRIPTION:
There are three primary objectives to the study: (1) Determine which dimensions of e-cigarette product diversity differentially affect product appeal in the overall population of tobacco product users as well as affect product appeal across young adult e-cigarette users and middle-age/older adult smokers; (2) Determine which dimensions of e-cigarette product diversity differentially affect product appeal in the overall population of tobacco product users as well as affect abuse liability in young adult e-cigarette users and the ability to resist smoking in adult smokers; (3) Determine the affect of product characteristics on e-cigarette nicotine delivery profile.

ELIGIBILITY:
Inclusion Criteria:

Vapers/E-cigarette Users

* Regular use of e-cigarettes/vaping devices containing nicotine

Cigarette Smokers

- Regular use of cigarettes containing nicotine

Exclusion Criteria:

* Pregnant or planning to become pregnant

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Subjective Appeal Rating Measure | 1 hour
  This self-report measures of subjective product appeal will be completed following e-cigarette self-administration and review of marketing strategies. Scores can range from 0 to 100 for the appeal rating, with lower scores representing lower levels of appeal and higher scores representing higher levels of appeal.
Sensory Attributes | 1 hour
  Self-report measures of product sensory attributes will be completed following e-cigarette self-administration and review of marketing strategies. Scores can range from 0 to 100 for the sensory attribute rating, with lower scores representing lower levels of liking the sensory attribute and higher scores representing greater liking of the sensory attribute.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No